CLINICAL TRIAL: NCT03552757
Title: Effect and Safety of Semaglutide 2.4 mg Once-weekly in Subjects With Overweight or Obesity and Type 2 Diabetes
Brief Title: Research Study Investigating How Well Semaglutide Works in People With Type 2 Diabetes Suffering From Overweight or Obesity
Acronym: STEP 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4374; U1111-1200-8148 (Other: World Health Organization (WHO)); 2017-003414-10 (Other: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Semaglutide 1.0 mg (Experimental): Participants will receive semaglutide 1.0 mg and semaglutide placebo I during 68-week treatment period in addition to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Semaglutide 1.0 mg; Drug: Placebo I (Semaglutide)
- Semaglutide 2.4 mg (Experimental): Participants will receive semaglutide 2.4 mg and semaglutide placebo II during 68-week treatment period in addition to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Semaglutide 2.4 mg; Drug: Placebo II (Semaglutide)
- Semaglutide placebo I/II (Placebo Comparator): Participants will receive semaglutide placebo I and II during 68-week treatment period in addition to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Placebo I (Semaglutide); Drug: Placebo II (Semaglutide)

INTERVENTIONS:
Drug: Semaglutide 1.0 mg — Subcutaneous (s.c.) injections of semaglutide once weekly at an escalating doses (0.25 mg/week, 0.5 mg/week, 1.0 mg mg/week). The dose will be escalated to next level every 4 weeks.
  Arms: Semaglutide 1.0 mg
Drug: Semaglutide 2.4 mg — Subcutaneous injections of semaglutide once weekly at an escalating doses (0.25 mg/week, 0.5 mg/week, 1.0 mg mg/week, 1.7 mg/week and 2.4 mg/week). The dose will be escalated to next level every 4 weeks.
  Arms: Semaglutide 2.4 mg
Drug: Placebo I (Semaglutide) — S.c. injections of placebo once weekly at a similar dose escalation manner as semaglutide 2.4 mg (placebo matched to semaglutide 0.25 mg/week, 0.5 mg/week, 1.0 mg mg/week, 1.7 mg/week and 2.4 mg/week). The dose will be escalated to next level every 4 weeks.
  Arms: Semaglutide 1.0 mg; Semaglutide placebo I/II
Drug: Placebo II (Semaglutide) — S.c. injections of placebo once weekly at a similar dose escalation manner as semaglutide 1.0 mg (placebo matched to semaglutide 0.25 mg/week, 0.5 mg/week, 1.0 mg mg/week). The dose will be escalated to next level every 4 weeks.
  Arms: Semaglutide 2.4 mg; Semaglutide placebo I/II

SUMMARY:
This study will look at the change in the participant's body weight from the start to the end of the study. This is to compare the effect on body weight in people taking semaglutide (a new medicine) and people taking "dummy" medicine. In addition to taking the study medicine, the participant will have talks with study staff about healthy food choices, how to be more physically active and what else the participant can do to lose weight. Overweight and obesity is associated with an increased risk of type 2 diabetes. Therefore, weight loss has shown to have a beneficial impact on the blood sugar levels. The participant will either get semaglutide or "dummy" medicine - which treatment the participant get is decided by chance. The participant will need to take 2 injections at the same time once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. The study will last for about 1.5 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Body Mass Index (BMI) greater than or equal to 27 kg/m^2 '
* History of at least one self-reported unsuccessful dietary effort to lose body weight
* Diagnosed with type 2 diabetes (haemoglobin A1c 7-10% (53-86 mmol/mol) (both inclusive)) 180 days or longer prior to the day of screening

Exclusion Criteria:

* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of less than 30 mL/min/1.73 m^2 (less than 60 ml/min/1.73 m^2 in subjects treated with Sodium-glucose Cotransporter 2 Inhibitors) according to chronic kidney disease (CKD)-Epidemiology Collaboration (EPI) creatinine equation as defined by Kidney Disease: Improving Global Outcomes (KDIGO) 2012 by the central laboratory at screening
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or an equally qualified health care provider (e.g. optometrist) within the past 90 days prior to screening or in the period between screening and randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1210 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (120):
- United States (45):
  - Novo Nordisk Investigational Site, Buena Park, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Alpharetta, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, West Des Moines, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Olive Branch, Mississippi
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Hickory, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Shavano Park, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
- Argentina (5):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Chacabuco
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mendoza
  - Novo Nordisk Investigational Site, Santiago del Estero
- Canada (8):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Stoney Creek, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Saint-Marc-des-Carrieres, Quebec
- Germany (8):
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Lingen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Schweinfurt
  - Novo Nordisk Investigational Site, Stuttgart
- Greece (3):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Haidari-Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- India (12):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Secunderabad
- Japan (10):
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Mitaka-shi, Tokyo
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Tochigi
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (4):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tomsk
- South Africa (4):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
- Spain (7):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, San Cristóbal de La Laguna
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valladolid
- United Arab Emirates (3):
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Hatta
  - Novo Nordisk Investigational Site, Umm Al Quwain City
- United Kingdom (10):
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Crewe
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Harrogate, North Yorkshire
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Soham
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Watford
  - Novo Nordisk Investigational Site, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com

REFERENCES:
- [Background] Kushner RF, Calanna S, Davies M, Dicker D, Garvey WT, Goldman B, Lingvay I, Thomsen M, Wadden TA, Wharton S, Wilding JPH, Rubino D. Semaglutide 2.4 mg for the Treatment of Obesity: Key Elements of the STEP Trials 1 to 5. Obesity (Silver Spring). 2020 Jun;28(6):1050-1061. doi: 10.1002/oby.22794. PMID 32441473
- [Result] Davies M, Faerch L, Jeppesen OK, Pakseresht A, Pedersen SD, Perreault L, Rosenstock J, Shimomura I, Viljoen A, Wadden TA, Lingvay I; STEP 2 Study Group. Semaglutide 2.4 mg once a week in adults with overweight or obesity, and type 2 diabetes (STEP 2): a randomised, double-blind, double-dummy, placebo-controlled, phase 3 trial. Lancet. 2021 Mar 13;397(10278):971-984. doi: 10.1016/S0140-6736(21)00213-0. Epub 2021 Mar 2. PMID 33667417
- [Derived] Schattenberg JM, Gronbaek H, Kliers I, Ladelund S, Long MT, Nygard SB, Sanyal AJ, Davies MJ. Proteomic signatures reflect effects of semaglutide treatment for MASH. JHEP Rep. 2025 Jul 22;7(10):101521. doi: 10.1016/j.jhepr.2025.101521. eCollection 2025 Oct. PMID 40980163
- [Derived] Wadden TA, Brown GK, Egebjerg C, Frenkel O, Goldman B, Kushner RF, McGowan B, Overvad M, Fink-Jensen A. Psychiatric Safety of Semaglutide for Weight Management in People Without Known Major Psychopathology: Post Hoc Analysis of the STEP 1, 2, 3, and 5 Trials. JAMA Intern Med. 2024 Nov 1;184(11):1290-1300. doi: 10.1001/jamainternmed.2024.4346. PMID 39226070
- [Derived] Heerspink HJL, Apperloo E, Davies M, Dicker D, Kandler K, Rosenstock J, Sorrig R, Lawson J, Zeuthen N, Cherney D. Effects of Semaglutide on Albuminuria and Kidney Function in People With Overweight or Obesity With or Without Type 2 Diabetes: Exploratory Analysis From the STEP 1, 2, and 3 Trials. Diabetes Care. 2023 Apr 1;46(4):801-810. doi: 10.2337/dc22-1889. PMID 36801984
- [Derived] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 149 sites in 12 countries as follows: Argentina (5 sites), Canada (10 sites), Germany (9 sites), Greece (6 sites), India (18 sites), Japan (12 sites), Russian Federation (9 sites), South Africa (6 sites), Spain (8 sites), United Arab Emirates (5 sites), United Kingdom (10 sites) and United States (51 sites).
Pre-assignment Details: Participants were randomised in 1:1:1 ratio to receive either 'semaglutide 2.4 milligram (mg) and placebo II (placebo matched to semaglutide 1.0 mg) once weekly', 'semaglutide 1.0 mg and placebo I (placebo matched to semaglutide 2.4 mg) once weekly' or 'placebo I and placebo II once weekly'.
Groups:
- Semaglutide 1.0 mg: Participants received once-weekly subcutaneous (s.c; under the skin) semaglutide injections for 68 weeks: 0.25 mg from week 1-4, 0.5 mg from week 5-8 and 1.0 mg from week 9-68. Participants also received once-weekly placebo I (placebo matched to semaglutide 2.4 mg) s.c. injection for 68 weeks. Participants received the treatments as an adjunct to a reduced calorie diet and increased physical activity.
- Semaglutide 2.4 mg: Participants received once-weekly s.c semaglutide injections for 68 weeks: 0.25 mg from week 1-4, 0.5 mg from week 5-8, 1.0 mg from week 9-12, 1.7 mg from week 13-16 and 2.4 mg from week 17-68. Participants also received once-weekly placebo II (placebo matched to semaglutide 1.0 mg) s.c. injection for 68 weeks. Participants received the treatments as an adjunct to a reduced calorie diet and increased physical activity.
- Placebo: Participants received once-weekly s.c placebo injections (both placebo I (placebo matched to semaglutide 1.0 mg) and placebo II (placebo matched to semaglutide 2.4 mg) for 68 weeks. Participants received the treatments as an adjunct to a reduced calorie diet and increased physical activity.
Period: Overall Study
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Started | 403 | 404 | 403
Exposed | 402 | 403 | 402
Full Analysis Set (FAS) | 403 | 404 | 403
Safety Analysis Set (SAS) | 402 | 403 | 402
Completed | 390 | 391 | 383
Not Completed | 13 | 13 | 20
Not completed — Withdrawal by Subject | 10 | 5 | 12
Not completed — Lost to Follow-up | 2 | 7 | 7
Not completed — Death | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) which comprised all randomised participants.
Groups:
- Semaglutide 1.0 mg: Participants received once-weekly s.c semaglutide injections for 68 weeks: 0.25 mg from week 1-4, 0.5 mg from week 5-8 and 1.0 mg from week 9-68. Participants also received once-weekly placebo I (placebo matched to semaglutide 2.4 mg) s.c. injection for 68 weeks. Participants received the treatments as an adjunct to a reduced calorie diet and increased physical activity.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 403 | 404 | 403 | 1210
Age, Continuous [Mean (Standard Deviation); unit: Year] | 56 (10) | 55 (11) | 55 (11) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 223 | 190 | 616
  Male | 200 | 181 | 213 | 594
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 272 | 237 | 242 | 751
  Asian | 97 | 112 | 108 | 317
  Black or African American | 28 | 35 | 37 | 100
  Other | 6 | 16 | 13 | 35
  American Indian or Alaska Native | 0 | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Not Applicable | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 344 | 357 | 354 | 1055
  Hispanic or Latino | 59 | 47 | 49 | 155
  Not Applicable | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%) - Semaglutide 2.4 mg Versus Placebo
Description: Change in body weight (%) from baseline (week 0) to week 68 is presented. Results are based on the data from both in-trial and on-treatment observation periods. In-trial observation period: the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact (week 75). On-treatment observation period: the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 2-week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0) to week 68
Population: Overall number of participants analysed = FAS which comprised all randomised participants. Number analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of body weight
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 404 | 403
Percentage point of body weight
  In-trial observation period: number analyzed (Participants) | 388 | 376
  In-trial observation period | -9.9 (8.0) | -3.3 (5.5)
  On-treatment observation period: number analyzed (Participants) | 351 | 340
  On-treatment observation period | -10.7 (7.8) | -3.1 (5.2)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Results are based on the data from in-trial observation period. Week 68 responses were analysed using an analysis of covariance model (ANCOVA) with randomised treatment, stratification groups (oral anti-diabetic (OAD) treatment status and HbA1c category at screening) and the interaction between stratification groups as factors and baseline body weight as covariate; Test type: Superiority; p < 0.0001, ANCOVA; Treatment difference = -6.21, 95% CI 2-sided [-7.28 to -5.15]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Results are based on the data from on-treatment observation period. All responses prior to first discontinuation of treatment (or initiation of other anti-obesity medication or bariatric surgery) were included in a mixed model for repeated measurements (MMRM) with randomised treatment, stratification groups (OAD treatment status and HbA1c category at screening) and the interaction between stratification groups as factors and baseline body weight as covariate, all nested within visit; Test type: Superiority; p < 0.0001, MMRM; Treatment difference = -7.57, 95% CI 2-sided [-8.56 to -6.58]

2. Primary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥5% - Semaglutide 2.4 mg Versus Placebo
Description: Number of participants who achieved weight reduction ≥5% of their baseline body weight (yes/no) at week 68 is presented. Results are based on the data from both in-trial and on-treatment observation periods. In-trial observation period: the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact. On-treatment observation period: the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 2 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: At week 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 404 | 403
Participants
  In-trial observation period: number analyzed (Participants) | 388 | 376
  In-trial observation period: Yes | 267 | 107
  In-trial observation period: No | 121 | 269
  On-treatment observation period: number analyzed (Participants) | 351 | 340
  On-treatment observation period: Yes | 257 | 94
  On-treatment observation period: No | 94 | 246
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Results are based on the data from in-trial observation period. Week 68 responses were analysed using a binary logistic regression model with randomised treatment, stratification groups (OAD treatment status and HbA1c category at screening) and the interaction between stratification groups as factors and baseline body weight as covariate; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.88, 95% CI 2-sided [3.58 to 6.64]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Results are based on the data from on-treatment observation period. All responses prior to first discontinuation of treatment (or initiation of other anti-obesity medication or bariatric surgery) were included in a MMRM with randomised treatment, stratification groups (OAD treatment status and HbA1c category at screening) and the interaction between stratification groups as factors and baseline body weight as covariate, all nested within visit; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 8.69, 95% CI 2-sided [6.31 to 11.97]

3. Secondary Outcome: Change in Body Weight (%) - Semaglutide 2.4 mg Versus Semaglutide 1.0 mg
Description: Change in body weight (%) from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of body weight
Arm/Group | Semaglutide 2.4 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 388 | 380
Percentage point of body weight | -9.9 (8.0) | -7.2 (6.6)

4. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥5% - Semaglutide 2.4 mg Versus Semaglutide 1.0 mg
Description: Number of participants who achieved weight reduction ≥5% of their baseline body weight (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 388 | 380
Participants
  Yes | 267 | 217
  No | 121 | 163

5. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimetre (cm)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 380 | 387 | 375
Centimetre (cm) | -6.9 (6.8) | -9.7 (8.1) | -4.3 (6.5)

6. Secondary Outcome: Change in Body Weight (Kg)
Description: Change in body weight (kg) from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 380 | 388 | 376
Kilogram (kg) | -7.1 (6.7) | -9.9 (8.5) | -3.4 (6.2)

7. Secondary Outcome: Change in BMI
Description: Change in body mass index (BMI) from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 380 | 388 | 376
kilogram per square meter (kg/m^2) | -2.6 (2.4) | -3.6 (3.1) | -1.2 (2.1)

8. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥10%
Description: Number of participants who achieved weight reduction ≥10% of their baseline body weight (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 380 | 388 | 376
Participants
  Yes | 109 | 177 | 31
  No | 271 | 211 | 345

9. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥15%
Description: Number of participants who achieved weight reduction ≥15% of their baseline body weight (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 380 | 388 | 376
Participants
  Yes | 52 | 100 | 12
  No | 328 | 288 | 364

10. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥20%
Description: Number of participants who achieved weight reduction ≥20% of their baseline body weight (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 380 | 388 | 376
Participants
  Yes | 18 | 51 | 6
  No | 362 | 337 | 370

11. Secondary Outcome: Change in HbA1c (%)
Description: Change in glycated haemoglobin (HbA1c (%)) from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 376 | 381 | 374
Percentage point of HbA1c | -1.5 (1.1) | -1.7 (1.2) | -0.3 (1.3)

12. Secondary Outcome: Change in HbA1c (mmol/Mol)
Description: Change in HbA1c (mmol/mol) from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: millimoles per mole (mmol/mol)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 376 | 381 | 374
millimoles per mole (mmol/mol) | -16.9 (12.3) | -18.7 (13.0) | -3.4 (14.3)

13. Secondary Outcome: Change in FPG (mg/dL)
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 367 | 375 | 370
milligrams per deciliter (mg/dL) | -36.5 (45.1) | -37.9 (45.9) | -2.3 (53.1)

14. Secondary Outcome: Change in Fasting Serum Insulin
Description: Change in fasting serum insulin from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles per litre (pmol/L)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 352 | 360 | 351
Picomoles per litre (pmol/L) | 0.94 (59.8) | 0.90 (65.4) | 0.93 (53.6)

15. Secondary Outcome: Participants Who Achieve (Yes/no): HbA1c <7.0% (53 mmol/Mol)
Description: Number of participants who achieved HbA1c <7% (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 376 | 381 | 374
Participants
  Yes | 272 | 299 | 99
  No | 104 | 82 | 275

16. Secondary Outcome: Participants Who Achieve (Yes/no): HbA1c ≤6.5% (48 mmol/Mol)
Description: Number of participants who achieved HbA1c ≤6.5% (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 376 | 381 | 374
Participants
  Yes | 226 | 257 | 58
  No | 150 | 124 | 316

17. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥10% and HbA1c <7.0%
Description: Number of participants who achieved weight reduction ≥10% of their baseline body weight and HbA1c <7.0% (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 376 | 381 | 374
Participants
  Yes | 105 | 170 | 25
  No | 271 | 211 | 349

18. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction ≥15% and HbA1c <7.0%
Description: Number of participants who achieved weight reduction ≥15% of their baseline body weight and HbA1c <7.0% (yes/no) at week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 376 | 381 | 374
Participants
  Yes | 49 | 98 | 11
  No | 327 | 283 | 363

19. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 379 | 387 | 376
Millimetre of mercury (mmHg) | -3 (15) | -4 (14) | 0 (15)

20. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to week 68 is presented. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 379 | 387 | 376
Millimetre of mercury (mmHg) | -1 (9) | -2 (9) | -1 (9)

21. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol (measured in milligram per decilitre (mg/dL)) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 380 | 373
Ratio of total cholesterol | 0.97 (20.1) | 0.99 (17.9) | 1.00 (18.9)

22. Secondary Outcome: Change in HDL Cholesterol
Description: Change in high density lipoprotein (HDL; measured in mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 375 | 369
Ratio of HDL cholesterol | 1.06 (16.0) | 1.07 (15.7) | 1.04 (15.3)

23. Secondary Outcome: Change in LDL Cholesterol
Description: Change in low density lipoprotein (LDL; measured in mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 380 | 373
Ratio of LDL cholesterol | 0.99 (37.5) | 1.00 (30.9) | 1.00 (28.9)

24. Secondary Outcome: Change in VLDL Cholesterol
Description: Change in very low density lipoprotein (VLDL; measured in mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 380 | 373
Ratio of VLDL cholesterol | 0.82 (42.1) | 0.80 (42.0) | 0.92 (40.5)

25. Secondary Outcome: Change in Free Fatty Acids
Description: Change in free fatty acids (measured in mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 353 | 361 | 354
Ratio of free fatty acids | 0.85 (61.4) | 0.84 (68.7) | 1.01 (62.3)

26. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides (measured in mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 380 | 373
Ratio of triglycerides | 0.81 (44.5) | 0.79 (43.8) | 0.92 (44.5)

27. Secondary Outcome: Change in hsCRP
Description: Change in high sensitivity C-reactive protein (hsCRP; measured in milligram per ilitre (mg/L)) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 380 | 373
Ratio of hsCRP | 0.59 (115.7) | 0.50 (125.7) | 0.84 (90.9)

28. Secondary Outcome: Change in PAI-1 Activity
Description: Change in Plasminogen Activator Inhibitor-1 (PAI-1; measured in arbritary units per millilitre (AU/mL)) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of PAI-1 activity
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 334 | 353 | 336
Ratio of PAI-1 activity | 1.21 (73.7) | 1.06 (80.8) | 1.42 (68.9)

29. Secondary Outcome: Change in Short Form 36 v2.0 Acute (SF-36) (Physical Functioning Score)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint shows results for 'physical functioning domain'. The 0-100 scale scores from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively. Change from week 0 in the domain scores were evaluated at week 68. A positive change score indicates an improvement since baseline. Results are based on the data from in-trial observation period.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 370 | 376 | 365
Score on a scale | 2.1 (6.8) | 2.8 (7.7) | 0.8 (7.0)

30. Secondary Outcome: Change in SF-36 (All Scores Except Physical Functioning)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint shows results for all the domains, except physical functioning. The 0-100 scale scores from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively. Change from week 0 in the domain scores and component summary scores were evaluated at week 68. A positive change score indicates an improvement since baseline. Results are based on the data from in-trial observation period.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 370 | 376 | 365
Score on a scale
  Role-Physical | 0.6 (6.9) | 0.8 (7.4) | 0.0 (7.1)
  Bodily Pain | 0.4 (8.3) | 0.3 (9.0) | -0.4 (8.6)
  General Health | 1.7 (7.2) | 2.2 (7.3) | 0.6 (7.5)
  Vitality | -0.1 (7.8) | 0.8 (7.9) | -0.9 (7.9)
  Social Functioning | -0.3 (6.6) | 0.2 (6.6) | -0.7 (7.4)
  Role-Emotional | -0.4 (7.3) | -0.4 (7.7) | -1.1 (7.8)
  Mental Health | -0.9 (7.5) | -0.4 (6.9) | -1.6 (7.5)
  Physical component summary | 1.9 (6.4) | 2.3 (7.2) | 0.9 (6.6)
  Mental component summary | -1.4 (7.4) | -0.9 (6.9) | -1.8 (7.6)

31. Secondary Outcome: Change in IWQOL-Lite for CT (Physical Function Domain (5-items) Score)
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on patients' quality of life within the context of clinical trials. IWQOL-Lite-CT is a 20-item questionnaire-based instrument used to assess the impact of body weight changes on participant's overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning. This endpoint shows results for 'physical function domain'. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 369 | 376 | 365
Score on a scale | 8.5 (18.8) | 11.4 (20.8) | 4.9 (20.4)

32. Secondary Outcome: Change in IWQOL-Lite for CT (All Scores Except Physical Function)
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on patients' quality of life within the context of clinical trials. IWQOL-Lite-CT is a 20-item questionnaire-based instrument used to assess the impact of body weight changes on participant's overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning. This endpoint shows results for 'physical and psychosocial domains, and for total'. Results are based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 369 | 376 | 365
Score on a scale
  Physical | 7.6 (18.0) | 11.0 (19.6) | 4.4 (19.1)
  Psychosocial | 8.6 (15.7) | 9.6 (16.7) | 5.6 (16.5)
  Total | 8.2 (14.8) | 10.1 (15.9) | 5.2 (15.5)

33. Secondary Outcome: Participants Who Achieve (Yes/no): Responder Definition Value for SF-36 Physical Functioning Score
Description: The observed number of participants experiencing a meaningful within participant improvement in SF-36 Physical function after 68 weeks was determined based on two thresholds. The threshold of 4.3 is the default generic responder threshold defined in SF-36 manual for a general population. The threshold of 3.7 is specific for overweight or obese population included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on Food and Drug Administration (FDA) recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers number of participants who have not achieved an improvement in score greater than or equal to the threshold. Endpoint was evaluated based on in-trial observation period which is the uninterrupted time interval from randomization (week 0) to last trial related subject-site contact (week 75).
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 370 | 376 | 365
Participants
  Yes (with threshold 4.3) | 88 | 111 | 68
  No (with threshold 4.3) | 282 | 265 | 297
  Yes (with threshold 3.7) | 130 | 158 | 102
  No (with threshold 3.7) | 240 | 218 | 263

34. Secondary Outcome: Participants Who Achieve (Yes/no): Responder Definition Value for IWQOL-Lite for CT Physical Function Domain (5-items) Score
Description: The observed number of participants experiencing a meaningful within participant improvement in IWQOL-Lite-CT physical function after 68 weeks was determined based on two different thresholds. The threshold of 20 was a preliminary responder threshold based on earlier studies. The threshold of 14.6 is specific for the population with overweight or obesity included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on FDA recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers the number of participants who have not achieved an improvement in score greater than or equal to the threshold. The endpoint was evaluated based on the in-trial observation period which was defined as the uninterrupted time interval from randomization (week 0) to last trial related subject-site contact (week 75).
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 369 | 376 | 365
Participants
  Yes (with threshold 20) | 107 | 131 | 83
  No (with threshold 20) | 262 | 245 | 282
  Yes (with threshold 14.6) | 144 | 160 | 113
  No (with threshold 14.6) | 225 | 216 | 252

35. Secondary Outcome: Number of TEAEs - Semaglutide 2.4 mg Versus Placebo
Description: Adverse events (AEs) with onset during the on-treatment observation period were defined as treatment-emergent AEs (TEAEs). On-treatment observation period: the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least seven consecutive missed doses.
Time Frame: Week 0 to week 75
Population: Safety analysis set (SAS) included all randomised participants exposed to at least one dose of randomised treatment. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 403 | 402
Events | 2197 | 1388

36. Secondary Outcome: Number of SAEs - Semaglutide 2.4 mg Versus Placebo
Description: Serious adverse event (SAE) results are based on the on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least seven consecutive missed doses.
Time Frame: Week 0 to week 75
Population: SAS included all randomised participants exposed to at least one dose of randomised treatment. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 403 | 402
Events | 71 | 53

37. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemia Episodes - Semaglutide 2.4 mg Versus Placebo
Description: Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least 7 consecutive missed doses. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. plasma glucose (PG) concentrations may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG concentration. Blood glucose (BG) confirmed symptomatic hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0 to week 75
Population: as for outcome 36
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 403 | 402
Episodes | 51 | 18

38. Secondary Outcome: Change in Pulse - Semaglutide 2.4 mg Versus Placebo
Description: Change in pulse from baseline (week 0) to week 68 is presented. Results are based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 2 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 351 | 340
Beats/minute | 2 (9) | 0 (9)

39. Secondary Outcome: Change in Amylase - Semaglutide 2.4 mg Versus Placebo
Description: Change in amylase (units/litre) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 2 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 350 | 338
Ratio of amylase | 1.24 (28.3) | 1.06 (25.0)

40. Secondary Outcome: Change in Lipase - Semaglutide 2.4 mg Versus Placebo
Description: Change in lipase (units/litre) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 2 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 350 | 338
Ratio of lipase | 1.41 (57.2) | 0.99 (51.8)

41. Secondary Outcome: Change in Calcitonin - Semaglutide 2.4 mg Versus Placebo
Description: Change in calcitonin (nanogram/litre) from baseline (week 0) to week 68 is presented as ratio to baseline. Results are based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 2 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 348 | 339
Ratio of calcitonin | 0.94 (60.3) | 0.96 (38.6)

ADVERSE EVENTS:
Time Frame: Week 0 to week 75. Results are based on the SAS which included all randomised participants exposed to at least one dose of randomised treatment.
Description: All presented AEs are treatment-emergent (i.e., TEAEs).
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/402 | 1/403 | 1/402
Serious Adverse Events (participants affected / at risk) | 31/402 | 40/403 | 37/402
Other Adverse Events (participants affected / at risk) | 261/402 | 284/403 | 190/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=402) | Semaglutide 2.4 mg (N=403) | Placebo (N=402)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Cerebral artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sperm aspiration (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=402) | Semaglutide 2.4 mg (N=403) | Placebo (N=402)
Abdominal distension (Gastrointestinal disorders) | 9 (12) | 24 (30) | 11 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (27) | 23 (29) | 20 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (30) | 27 (30) | 14 (15)
Constipation (Gastrointestinal disorders) | 51 (70) | 70 (82) | 22 (26)
Decreased appetite (Metabolism and nutrition disorders) | 29 (33) | 38 (41) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 88 (157) | 86 (141) | 48 (66)
Dyspepsia (Gastrointestinal disorders) | 27 (27) | 25 (30) | 5 (5)
Fatigue (General disorders) | 19 (26) | 28 (29) | 4 (4)
Flatulence (Gastrointestinal disorders) | 21 (25) | 16 (21) | 7 (9)
Gastroenteritis (Infections and infestations) | 21 (25) | 11 (12) | 12 (14)
Headache (Nervous system disorders) | 33 (48) | 31 (40) | 20 (27)
Nasopharyngitis (Infections and infestations) | 47 (69) | 68 (115) | 59 (92)
Nausea (Gastrointestinal disorders) | 128 (196) | 135 (248) | 37 (45)
Upper respiratory tract infection (Infections and infestations) | 37 (54) | 42 (48) | 38 (50)
Vomiting (Gastrointestinal disorders) | 54 (93) | 86 (186) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03552757/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03552757/SAP_003.pdf